CLINICAL TRIAL: NCT02744859
Title: Do Warning Labels Decrease Soda Purchasing?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Leslie John, Principal Investigator, Harvard University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB16-0222
Record Dates: First submitted 2016-04-13; First posted 2016-04-20 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Decision Making; Consumption; Economics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Calorie Label (Experimental): Labels will read "[lower calorie bound] - [upper calorie bound] calories per container. 2,000 calories a day is used for general nutrition advice but calorie needs vary."
  Interventions: Other: Label Condition
- Warning Label (Experimental): Labels will read "WARNING: Drinking beverages with added sugar(s) contributes to obesity, diabetes, and tooth decay."
  Interventions: Other: Label Condition
- Warning Label with Graphics (Experimental): Labels will read "WARNING: Drinking beverages with added sugar(s) contributes to obesity, diabetes, and tooth decay." These labels will also have graphic depictions of each health condition above the corresponding text.
  Interventions: Other: Label Condition
- No label (No Intervention): We will also have a condition where no labels are presented-- business as usual.

INTERVENTIONS:
Other: Label Condition — Labels will be presented in front of drinks. We will vary the messaging presented to the consumer.
  Arms: Calorie Label; Warning Label; Warning Label with Graphics

SUMMARY:
Investigators will run a field study evaluating the impact different labels have on the purchasing of sugar sweetened beverages. This field study will take place in a hospital cafeteria.

DETAILED DESCRIPTION:
In a hospital cafeteria investigators will label all sugar sweetened beverages to evaluate their impact on purchasing.

Investigators will collect baseline data for two weeks on beverage sales at the hospital cafe. Following this data collection investigators will introduce a calorie label which reads "Each beverage contains [lower calorie bound]-[upper calorie bound] calories per container. 2,000 calories a day is used for general nutrition advice but calorie needs vary." These signs will be posted for two weeks and investigators will collect sales data. Following this intervention investigators will remove the signs and collect sales data for two weeks. At the end of this no label period, investigators will introduce the second intervention, a warning label. This label will read "WARNING: Drinking beverages with added sugar(s) contributes to obesity, diabetes, and tooth decay." This label will also be posted for two weeks and investigators will collect sales data. Investigators will then remove these signs and collect sales data for two weeks. Finally, investigators will introduce the third intervention: a warning label with graphic labels. This label will read "WARNING: Drinking beverages with added sugar(s) contributes to obesity, diabetes and tooth decay." However this sign will also include a visual depiction of each health consequence. Investigators will collect sales data for this two week period. After this intervention investigators will collect sales data for an additional two weeks and then administer a brief survey to cafeteria customers to better understand their impressions of the labels.

ELIGIBILITY:
Inclusion Criteria:

* Customers of the hospital cafeteria.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6000 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Sweetened beverages purchased | 2 week condition blocks
  We will sum the total number of sugar sweetened beverages sold in each condition using the Universal Product Code (UPC) for bottled beverages and syrup weight for fountain beverages.

SECONDARY OUTCOMES:
Unsweetened beverages purchased | 2 week condition blocks
  We will sum the total number of unsweetened beverages sold in each condition using the Universal Product Code (UPC) for bottled beverages and syrup weight for fountain beverages.
Beverage calories sold | 2 week condition blocks
  We will calculate the number of beverage calories sold during each condition, using the Universal Product Code (UPC) for bottled beverages, syrup weight for fountain beverages, and the products' nutritional information.
Changes in types of beverages purchased | 2 week condition blocks
  We will examine any changes in the types of beverages purchased during each condition, using the Universal Product Code (UPC) for bottled beverages and syrup weight for fountain beverages. For example, if sugar-sweetened beverages sales decrease, do purchases of water increase?

CONTACTS AND LOCATIONS:
Overall Officials: Grant E Donnelly, MA, Principal Investigator — Harvard University; Laura Y Zatz, MPH, Principal Investigator — Harvard School of Public Health (HSPH)

REFERENCES:
- [Derived] Donnelly GE, Zatz LY, Svirsky D, John LK. The Effect of Graphic Warnings on Sugary-Drink Purchasing. Psychol Sci. 2018 Aug;29(8):1321-1333. doi: 10.1177/0956797618766361. Epub 2018 Jun 18. PMID 29912624